CLINICAL TRIAL: NCT00755924
Title: Prospective Randomized Clinical Trial Evaluating the Impact of Vinegar on High Density Lipoprotein
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Dr. Carmello Panetta, Park Nicollet Heart and Vascular Center/Park Nicollet Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 03635-07-C
Record Dates: First submitted 2008-09-17; First posted 2008-09-19 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2010-08

CONDITIONS: Cholesterol, HDL
MeSH Terms: interventions — Acetic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Vinegar — Apple cider vinegar 2 TBlsp/day
Other: Placebo — Water placebo colored with balsamic vinegar

SUMMARY:
This is a double-blinded randomized placebo controlled prospective clinical trial evaluating the impact of apple cider vinegar on serum HDL. 112 participants will be randomized to consume either 2 tablespoons of vinegar daily or a placebo containing a 2% balsamic vinegar solution in water. Baseline, two month and 4 month blood samples will be obtained for fasting lipids. The primary endpoint is met if HDL levels increase in the treatment arm versus baseline after 2 month intervention.

ELIGIBILITY:
Inclusion Criteria:

* Those older than 18 years of age
* Park Nicollet Health Services patient

Exclusion Criteria:

* Because of a potential positive effect of vinegar on improving diabetes mellitus8 and the subsequent change in medication regime for diabetes diabetic patients will be excluded from this study. If this study finds that vinegar does increase HDL levels, a subsequent study of diabetic patients will be conducted.
* History of allergy to apple cider vinegar
* Those with a terminal illness
* Diagnosis of Inflammatory bowel disease
* Those with Immunosuppression diseases
* Patients on dialysis
* Severe psychiatric illness who are unable to consent or reliably participate
* No evidence of end stage renal disease
* Those who use alcohol greater than or equal to 2 drinks per day
* Those who take in >3 tsp vinegar/day supplement
* Plans to increase exercise or begin diet during the protocol period
* Any use of niacin or niacin-like compounds
* Initiation of niacin, fibrates (eg gemfibrozil); statin or ezetimibe medication within the last 6 weeks or during the trial
* Inability to read English
* Age less than 18 years given clinical events would be unlikely in this population
* LDL greater than 160mg/dL and requires adjustment or addition of statin therapy (which could reduce HDL)
* History of liver failure in medical history review
* Current smoking (as this can reduce HDL levels and it would be unethical to require people to continue smoking during the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2008-06; Primary Completion 2009-08 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Change in HDL-Cholesterol level | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Park Nicollet Health Services, Minneapolis, Minnesota, United States